CLINICAL TRIAL: NCT06503068
Title: NAFLD Stigma vs MAFLD Stigma and Their Impact on Quality of Life in Egyptian Patients: A Survey Study
Brief Title: Impact of NAFLD vs MAFLD Stigma on Quality of Life in Egyptian Patients
Status: Recruiting | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Rania Mamdouh Elkafoury, Principle Investigator, Tanta University
Other Study IDs: 36264PR627/4/24
Record Dates: First submitted 2024-07-01; First posted 2024-07-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: NAFLD
Keywords: Metabolic- associated fatty liver disease (MAFLD); Non-alcoholic fatty liver disease (NAFLD); stigma; Metabolic dysfunction-associated steatotic liver disease (MASLD)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Social Stigma | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NAFLD/NASH patients: Patients ≥ 18 years old diagnosed with NAFLD/ NASH and willing to complete the survey.
  Interventions: Other: Questionnaire
- Physicians: Physicians treating patients with NAFLD/NASH (hepatologists, gastroenterologists, endocrinologists, and internal medicine physicians).
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — A questionnaire in both digital and written forms in both Arabic and English versions.

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) has become the leading cause of liver disease worldwide. The global burden of NAFLD is about 30% of the population, With a higher prevalence in Egypt about 47.5 %. The prevalence increases significantly with the presence of type 2 diabetes and obesity.

NAFLD is commonly associated with metabolic dysfunction and the development of cardiovascular disease. However, the NAFLD definition excludes other causes. It is not correlated with metabolic dysfunction and cardiovascular risk, so in 2020, the term metabolic-dysfunction-associated fatty liver disease (MAFLD) was suggested to replace the term NAFLD.

The nomenclature change was partly related to the stigma associated with the term NAFLD. As the words "alcoholic" and "fatty" were considered stigmatizing. A recent global survey showed that 26% of patients (57% in the USA and 7% in MENA) felt stigmatized relating to overweight/obesity and 8% of patients (22 % in the USA and 3% in MENA) felt stigmatized by the term NAFLD. While 34% and 38% of physicians considered the words "non-alcoholic" and "fatty" stigmatizing, respectively.

There is a discrepancy between the different regions of the world and between patients and providers regarding the perception of NAFLD/ MAFLD stigma. This study aims to assess the perception and stigmatization of various diagnostic terms (fatty liver, NAFLD & MAFLD) among Egyptian patients and physicians. Also, to assess the impact of stigma on the quality of life and the motivations and barriers for lifestyle modification which is the cornerstone of NAFLD/MAFLD management.

DETAILED DESCRIPTION:
This cross-sectional study will be carried out in collaboration between the Tropical Medicine Department and Public Health Department, Tanta University Hospitals. A questionnaire in both digital and written forms targeting patients with NAFLD/NASH and physicians treating NAFLD/NASH patients in Egypt.

Type of study:

Prospective, cross-sectional survey.

Duration of study:

Study will be carried out from May 2024 to August 2024 or until the target number is reached (about 500 subjects).

Target subjects:

The questionnaire will target a convenience sample of NAFLD/NASH patients and physicians treating NAFLD/NASH patients (about 500 subjects).

The questionnaire will be written and digital in both Arabic and English versions.

Methodology:

After designing the questionnaire, it will be discussed with other experts in the field, validity and reliability will be assessed and a pilot study will be done.

After an informed consent subject will answer a designed questionnaire either written or digital. 2 phases will be done The questionnaire will be divided into 3 sectors Sector 1: Demographic data: questions about [age, sex, residence, educational level, occupation (subspecialty), workplace] for all participants.

Sector 2: Socioeconomic level determination mainly for population :( Socio-economic data will be gathered through questions asking about the number of family members, number of rooms in the apartment, level of education, occupation, and cost per month).

Sector 3: the main work includes questions for patients: (patient awareness of NAFLD before diagnosis, presence and severity of liver fibrosis, presence of comorbidities, the diagnostic term they use to describe their disease, have they disclosed their condition to family or friends, have they experienced stigmatization or discriminations due to their disease and how frequently, how they feel about the words fatty, alcoholic, and metabolic, have they avoided or missed a visit with their physician due to NAFLD, patients concerns about the disease and its progression, barriers, and motivations for lifestyle modifications).

For physicians :(their clinical experience in NAFLD and the number of NAFLD/NASH patients they see per month, what terms they think are considered stigmatizing to their patients "fatty, non-alcoholic, overweight/obese, metabolic associated", does their patients feel discrimination due to their disease, would the name change help their patients, causes of frustration and discomfort when treating NAFLD patients, their opinion of what are the barriers and motivations for lifestyle modifications in their patients)

Ethical considerations:

A written or digital informed consent form authorizing the collection of this data was signed by all subjects The study will be approved by the Ethical Committee of Faculty of Medicine Tanta University.

The risks to the participants and measures needed to minimize these risks:

* The privacy of the data of the patients will be maintained.
* Any unexpected risks appear during the course of research will be cleared to the subjects and the ethical committee on time

Adequate provisions to maintain the privacy of participants and confidentially of data are as follows:

* A code number for each patient will be used, and symbols for the name and address will be kept in a special file.
* The investigators will hide the patients' names when the research is used
* The investigators will use the results of the research only for scientific aims and not use it in other aims.

The endpoint of this study:

Assess the prevalence of NAFLD/MAFLD stigma among both patients and physicians, and the beneficence of name change from NAFLD to MAFLD in Egypt to determine the factors leading to lifestyle modifications in NAFLD/MAFLD patients, thus improving patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old diagnosed with NAFLD/ NASH and willing to complete the survey.
* Physicians treating patients with NAFLD/NASH (hepatologists, gastroenterologists, endocrinologists, and internal medicine physicians).

Exclusion Criteria:

* Unwilling to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The questionnaire will target a convenience sample of NAFLD/NASH patients presenting to the Tropical Medicine Department clinics.
  physicians treating NAFLD/NASH patients in Egypt
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Awareness of NAFLD/MAFLD stigma in Egypt | till August 2024
  Using a questionnaire to assess awareness of stigma related to various diagnostic terms such as "fatty liver", "NAFLD", "MAFLD", and Metabolic dysfunction-associated steatotic liver disease "MASLD" in patients and in NAFLD/NASH treating physicians in Egypt.
Perception of NAFLD/MAFLD stigma in Egypt | till August 2024
  Using a questionnaire to assess perception of stigma related to various diagnostic terms such as "fatty liver", "NAFLD", "MAFLD", and "MASLD" in patients and in NAFLD/NASH treating physicians in Egypt.

SECONDARY OUTCOMES:
impact on quality of life | till August 2024
  Using a questionnaire to understand the impact of NAFLD vs MAFLD stigma on the quality of life in Egyptian patients
Motivations to lifestyle changes | till August 2024
  Using a questionnaire to evaluate the motivation for lifestyle changes in Egyptian patients
Barriers to lifestyle changes | till August 2024
  Using a questionnaire to evaluate the barriers for lifestyle changes in Egyptian patients

CONTACTS AND LOCATIONS:
Locations (1):
- Tropical medicine department, Tanta University Hospitals, Tanta, Gharbyea, Egypt